CLINICAL TRIAL: NCT06080971
Title: A Descriptive Study on Patterns of Persistent Neonatal Jaundice on Neonates and Children at Assiut University Children Hospital
Brief Title: Persistent Neonatal Jaundice on Neonates and Childern
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elham Allam Ahmed Abd elkarim, 71515,Assiut, Assiut University
Other Study IDs: persistent neonatal jaundice
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Describe demographic and clinical data of neonates & childern with (PNNJ) admitted to neonatology , hepatology & hematology units of Assiut university children hospital(AUCH).

Describe the distribution of etiologies of (PNNG) in neonates & children at AUCH.

Assess the outcome of (PNNJ) in neonates & childern admitted to AUCH .

DETAILED DESCRIPTION:
(persistent ) Prolonged neonatal jaundice (PNNJ)is defined as a serum bilirubin level higher than 85 μ mol/L (5 mg/dl) with yellowish discoloration of the skin ,sclera and conjunctiva , which persists at postnatal 14 days in full term infants and 21 days following the birth in preterm infants .

Etiologically it is important to distinguish jaundice type , is it unconjugated (indirect) or conjugated (direct)hyperbilirubinemia. A prolonged unconjugated hyperbilirubinemia is mostly caused by breastfeeding(which is the most common identified cause for prolonged unconjugated hyperbilirubinemia , It is known that breastmilk jaundice is seen at a rate of 1.3% in newborn infants and 2.4-25% in infants fed with breastmilk ) or to some pathological conditions such as hemolytic diseases (due to hereditary spherocytosis ,elliptocytosis or G6PD deficiency), congenital hypothyroidism, urinary infection, Crigler-Najjar or Gilbert syndromes ,pyloric stenosis ,sepsis.

Conjugated hyperbilirubinemia (Cholestatic jaundice ) is never physiologic. It affects 1/2,500 live births and it should be suspected in all jaundiced infants with light stools and dark urine , The differential diagnosis of cholestasis is extensive and a step-wise approach based on the initial history and physical examination is useful to rapidly identify the underlying etiology, Early recognition of neonatal cholestasis is essential to ensure timely treatment and optimal prognosis. (causes Include infections, anatomic abnormalities of the biliary system, endocrinopathies, genetic disorders ,cystic fibrosis, metabolic abnormalities, toxin and drug exposures, vascular abnormalities, neoplastic processes, and other miscellaneous causes , the most commonly identifiable causes are biliary atresia (BA) (25%-35%), genetic disorders (25%), metabolic diseases (20%), and a1-antitrypsin (A1AT) deficiency (10%) ; other pathological causes of prolonged conjugated hyperbilirubinemia are TORCH-S infections, Neonatal hepatitis syndrome, Choledochal cyst , Inspissated bile syndrome, Galactosemia ,Alagille syndrome & Hereditary bile acid synthesis disorders.

Diagnosis : is made according to the physical examination(skin ,stool & urine color, organomegaly) , clinical presentation , investigations &imaging findings.

The clinical presentation of(PNNJ) include yellowish discoloration of skin ,sclera &conjunctiva with change in color of stool &urine with or without organomegally persistent for more than 14 days in full term infants &21 days in preterm infants.

investigations: include CBC, serum total &direct Bilirubin , urine analysis &culture , Coombs' test, thyroid function tests, G6PD level, LFT, blood film, GAL1PUT, alpha - 1 antitrypsin test , screening for TORCH ,Ultrasonography of the abdomen.

Investigations for cholestatic jaundice :fine needle or true cut needle liver biopsy , magnetic resonance cholangiopacreatography (MRCP),endoscopic retrograde cholangiopancreatography (ERCP) and hepatobiliary scintigraphy.

Mortality/morbidity:

* Kernicterus or bilirubin encephalopathy, typically in infants It occurs when the unconjugated bilirubin levels cross 25 mg/dL in the blood it gets deposited in the brain tissue. The neurotoxicity leads to various neurologic sequelae as poor feeding ,irritability, a high-pitched cry ,no startle reflex ,lethargy , apnea , seizures ,cerebral palsy ,hearing loss ,learning disabilities.
* Liver cell failure &cirrhosis with portal hypertension are complications of neonatal cholestasis.

Treatment Phototherapy, intravenous immune globulin (IVIG), and exchange transfusion are the most widely used therapeutic modalities in certain instance as Gilbert syndrome medications as Phenobarbital an inducer of hepatic bilirubin metabolism a new therapy currently under development consist of inhibition of bilirubin production through blockage of heme oxygenase by using mesoporphyrins & protoporphyins .

Treatment of Cholestatic jaundice depend mainly on cause of cholestasis ,all neonates & children should receive fat soluble vitamins (A,K,E,D),surgical intervention (kasai procedure)or even liver transplantation may be done.

ELIGIBILITY:
Inclusion Criteria:

* All neonates and children with prolonged neonatal jaundice admitted to Neonatology , hepatology & hematology units at Assiut university children hospital through the period from 1/1/2024 to 31/12/2024.

Exclusion Criteria:

* Neonates with neonatal jaundice lasts less than 14 days in full term and 21 days in preterm infants

Ages: 14 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: neonates and children with prolonged neonatal jaundice
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-13 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Describe demographic and clinical data of neonates & childern with (PNNJ) admitted to neonatology , hepatology & hematology units of Assiut university children hospital(AUCH) Assess the outcome of (PNNJ) in neonates & childern admitted to AUCH . | Baseline
  Describe the distribution of etiologies of (PNNG) in neonates & children at AUCH.

REFERENCES:
- [Background] Siu SL, Chan LW, Kwong AN. Clinical and biochemical characteristics of infants with prolonged neonatal jaundice. Hong Kong Med J. 2018 Jun;24(3):270-276. doi: 10.12809/hkmj176990. Epub 2018 May 25. PMID 29807952
- [Background] Feldman AG, Sokol RJ. Neonatal Cholestasis. Neoreviews. 2013 Feb 1;14(2):10.1542/neo.14-2-e63. doi: 10.1542/neo.14-2-e63. PMID 24244109
- [Background] Moyer V, Freese DK, Whitington PF, Olson AD, Brewer F, Colletti RB, Heyman MB; North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. Guideline for the evaluation of cholestatic jaundice in infants: recommendations of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2004 Aug;39(2):115-28. doi: 10.1097/00005176-200408000-00001. PMID 15269615